CLINICAL TRIAL: NCT02109380
Title: The Impact of Short-term Bed-rest on Skeletal Muscle Mass and Insulin Sensitivity in Healthy, Young Men
Brief Title: Bed-rest, Muscle Mass and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Assistant Professor, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC 14-3-013
Record Dates: First submitted 2014-04-01; First posted 2014-04-09 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Disuse Atrophy
MeSH Terms: conditions — Muscular Disorders, Atrophic | interventions — Bed Rest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bed rest (Experimental): One week of bed rest.
  Interventions: Behavioral: Bed rest

INTERVENTIONS:
Behavioral: Bed rest

SUMMARY:
In the present study, the effects of 7 days of bed rest on muscle mass, muscle fiber characteristics and insulin sensitivity will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged from 18-35 years
* 18.5 < BMI < 30 kg/m2

Exclusion Criteria:

* Smoking
* Performing regular resistance training (3+ times per week, carrying out progressive training) in the previous 6 months
* Hypertension (according to WHO criteria) and/or cardiovascular disease
* Any back/leg/knee/neck/postural complaints
* Use of any prescribed medication
* Type 2 diabetes mellitus
* Any family history of thrombosis
* All co-morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthritis, spasticity/rigidity, all neurological disorders and paralysis).
* Myocardial infarction within the last 3 years
* Use of anti-coagulants

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps muscle cross-sectional area | One day before and directly after cessation of bed rest.

SECONDARY OUTCOMES:
Change in lower back cross-sectional area | One day before and directly after cessation of bed rest.
Change in leg and whole body lean tissue mass | One day before and directly after cessation of bed rest.
Change in muscle fiber size | One day before and directly after cessation of bed rest.
Change in muscle strength | One day before and directly after cessation of bed rest.
  Measured by 1-Repetition Maximum testing
Change in insulin sensitivity | One day before and directly after cessation of bed rest.
  Measured by hyperinsulinemic-euglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Dirks ML, Wall BT, van de Valk B, Holloway TM, Holloway GP, Chabowski A, Goossens GH, van Loon LJ. One Week of Bed Rest Leads to Substantial Muscle Atrophy and Induces Whole-Body Insulin Resistance in the Absence of Skeletal Muscle Lipid Accumulation. Diabetes. 2016 Oct;65(10):2862-75. doi: 10.2337/db15-1661. Epub 2016 Jun 29. PMID 27358494
- [Derived] Dirks ML, Backx EM, Wall BT, Verdijk LB, van Loon LJ. May bed rest cause greater muscle loss than limb immobilization? Acta Physiol (Oxf). 2016 Sep;218(1):10-2. doi: 10.1111/apha.12699. Epub 2016 May 20. No abstract available. PMID 27124248